CLINICAL TRIAL: NCT01172548
Title: A Multi-center, Single Arm, Phase II Study of Adjuvant Imatinib (Glivec®) in Patients Following the Resection of Primary Gastrointestinal Stromal Tumor ( GIST)
Brief Title: Safety and Efficacy Evaluation of Two Year Imatinib Treatment in Adjuvant Gastrointestinal Stromal Tumor (GIST)
Acronym: INV555
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSTI571BIC08
Record Dates: First submitted 2010-06-22; First posted 2010-07-29 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Resected GIST; primary GIST; tumor recurrence; KIT receptor; KIT positive; advanced GIST; minimal toxicity; GIST
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Recurrence | interventions — Imatinib Mesylate

ARMS (1):
- imatinib mesylate (Experimental)
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate
  Other Names: STI571; Gleevec/Glivec

SUMMARY:
GISTs are the most common mesenchymal tumors of the gastrointestinal tract. Approximately 95% of GISTs are positive for KIT (CD117)-the receptor for stem cell factor (SCF). GISTs are not responsive to conventional cytotoxic chemotherapy and disease often recurs even after complete resection with wide margins.

Imatinib mesylate (trade names: Glivec® and Gleevec®, imatinib, formerly STI571) is a signal transduction inhibitor targeting several protein-tyrosine kinases that are believed to play a role in the proliferation of tumor cells. In the Phase II study of imatinib [CSTI571B 2222] in 147 patients with recurrent or metastatic GIST, the partial response rates were 67% and 66% in patients treated at 400 mg/d and 600 mg/d, respectively. Skin rash and elevated transaminases were the most common reason for drug discontinuation. The most frequently reported AEs were mild nausea, vomiting, diarrhea, superficial edema (primarily periorbital or lower limb), myalgia and muscle cramps. Grade 3/4 events included fluid retention (pleural or pericardial effusions, ascites, and pulmonary edema), skin rash, liver toxicity and gastrointestinal (GI) hemorrhage. Myelosuppression (neutropenia and thrombocytopenia) was a consistent finding. Also, a tumor lysis-like syndrome occurred in some patients leading to gastrointestinal (GI) and/or intratumoral hemorrhage.

In a Phase 3, American College of Surgeons Oncology Group trial (ACOSOG Z9001) of adjuvant imatinib, imatinib significantly improved 1-year recurrence-free survival (RFS) compared with placebo.

In summary, clinical trials have shown that imatinib produces clinical benefit in most patients with unresectable or metastatic GIST and extends median survival from 19 to 57 months. Imatinib is the standard of care for advanced GIST and has received regulatory approval for the treatment of unresectable or metastatic GIST. Studies suggest that adjuvant imatinib for 1 year prolongs RFS in patients at high risk of recurrent disease and metastases following complete surgical resection of the primary GIST.

Imatinib is an appealing adjuvant therapy for resected GIST because:

1. Patients with primary GIST have a high chance of tumor recurrence
2. Conventional adjuvant treatment modalities are ineffective
3. Imatinib specifically inhibits the Kit receptor which is constitutively activated in most GISTs
4. Imatinib inhibits the growth of Kit positive cells in vitro
5. Imatinib is highly effective in many patients with advanced GIST in a Phase II trial
6. Imatinib has been associated with minimal toxicity in patients with advanced GIST and in patients with chronic myelogenous leukemia (CML)
7. Imatinib may have its greatest impact on survival when there is minimal disease.

Primary

* To assess Recurrence Free Survival Rate in patients with resected primary GIST who are treated with adjuvant imatinib for a duration of 2 years Secondary
* To compare Recurrence Free Survival, Overall Survival, and Time to Recurrence of patients with resected primary GIST who are treated with adjuvant imatinib for a duration of 2 years with historical data To assess the safety of imatinib given as adjuvant therapy for 2 years in patients with resected primary GIST

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of primary GIST (without peritoneal or distant metastasis) with positive immunostaining for KIT (CD117);
* Undergone complete gross resection of a primary GIST within 70 days prior to enrollment (includes R0 [negative microscopic margins] and R1 [positive microscopic margins]);
* Intermediate or high risk of recurrence based on Corless criteria (Section 5.1):

Exclusion Criteria:

* Patient has received prior therapy with imatinib, or any other molecular targeted or biological therapy.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2008-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Recurrence Free Survival Rate | 2 years

SECONDARY OUTCOMES:
Compare Recurrence Free Survival Rate to historical controls | 2 years
Compare Overall Survival to historical controls | 2 years
Compare Time To Recurrence to historical controls | 2 years
Adverse Events | 2 years
Treatment Compliance - tracking if the patient is coming to visits as per visit schedule in protocol | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- Novartis Investigative Site, Algiers, Algeria
- Egypt (2):
  - Novartis Investigative Site, Al Mansurah
  - Novartis Investigative Site, Cairo
- India (4):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, New Delhi
- Novartis Investigative Site, Amman, Jordan
- Novartis Investigative Site, Beirut, Lebanon
- Russia (6):
  - Novartis Investigative Site, Kazan', Tatarstan Republic
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Kursk
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Parktown, South Africa
- Taiwan (6):
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Lin-Ko
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Songkhla
- Novartis Investigative Site, Tunis, Tunisia
- Novartis Investigative Site, Ankara, Turkey (Türkiye)